CLINICAL TRIAL: NCT05345613
Title: Usage of Tranexamic Acid During Colonic Endoscopic Resection Procedures for Reduction Intraprocedural and Postprocedural Bleeding
Brief Title: Tranexamic Acid During Colonic Endoscopic Resection Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Anton Bermont, Doctor, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0017-22-ASF
Record Dates: First submitted 2022-04-10; First posted 2022-04-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid group (Experimental): standard solution for injection with TXA and without adrenaline
  Interventions: Drug: Tranexamic acid
- Standard therapy group (Placebo Comparator): standard solution for injection including adrenaline
  Interventions: Drug: Standard

INTERVENTIONS:
Drug: Tranexamic acid — Submucosal injection of standard solution including TXA during EMR procedure
  Other Names: TXA, Cyklokapron
  Arms: Tranexamic Acid group
Drug: Standard — Injection of standard solution
  Other Names: adrenaline, epinephrine
  Arms: Standard therapy group

SUMMARY:
Colonoscopy with polypectomy reduces the incidence and mortality associated with colon cancer. However, polypectomy is associated with adverse events such as bleeding. Tranexamic acid (TXA) is a synthetic derivative of lysine that exerts antifibrinolytic effects and may prevent bleeding. The investigators aim to evaluate the effect of local TXA on preventing intraprocedural and postprocedural bleeding in patients undergoing endoscopic mucosal resection (EMR) of large colon polyps.

DETAILED DESCRIPTION:
Endoscopic resection (ER) is an endoscopic technique used for the removal of sessile or flat neoplasms confined to the superficial layers (mucosa and submucosa) of the gastrointestinal (GI) tract.

This technique is not without risk, and clinically significant intraprocedural bleeding (CSIPB) and post-ER bleeding (CSPEB) remain the most frequently encountered serious adverse event.

The bleeding rate associated with ER varies for the different regions of the GI tract. This is most probably due to differences in the vascularity within the wall of the GI tract in each region.

For colonic ER, intraprocedural bleeding occurs in about 11% of cases with delayed bleeding up to 11%.

Management of CSIPB and CSPEB is often resource intensive and may necessitate hospitalization, blood transfusion, and repeat intervention. Some techniques, such as soft coagulation with the tip of a snare, epinephrine injection or hemoclip placement are used to decrease the risk of bleeding or treat active bleeding.

Diluted epinephrine, which causes vasoconstriction, is often added to the submucosal injection fluid because of the theoretical benefit of decreasing bleeding.

However, submucosal injection of epinephrine potentially can result in systemic effects such as severe hypertension, ventricular tachycardia, and intestinal ischemia.

Moreover, epinephrine injection may increase postprocedural pain and prolong patient observation after the procedure.

Tranexamic acid (TXA) is a synthetic derivative of lysine that exerts antifibrinolytic effects by inhibition of lysine binding sites on plasminogen molecules and therefore stabilizes the fibrin meshwork produced by secondary hemostasis. TXA was patented by Dr. S. Okamoto in 1957, and it was found to be significantly more potent than a precursor molecule known as epsilon-amino-caproic acid.

During the past few years, TXA has been 'rediscovered' and is currently used in many conditions that are associated with either overt or occult hemorrhage. It is one of the most frequently cited drugs in recent surgical publications involving nearly all surgical specialties.

After the CRASH-2 study which showed that administration of TXA to bleeding trauma patients within 3 hours of injury significantly reduced the risk of death due to bleeding and all-cause mortality without increasing the risk of vascular occlusive events, it has become an important part of trauma management.

It is also widely used in gynecological practice. Early treatment with TXA reduces death due to bleeding in women with post-partum hemorrhage, as well as total blood loss and transfusion requirements in hemorrhage after caesarean delivery. Therefore, TXA has been recommended by the WHO as part of postpartum hemorrhage management.

In gynecologic surgeries such as hysterectomy or myomectomy, the use of TXA significantly reduces blood loss without evidence of thrombotic events or deaths.

TXA is also commonly used in orthopedic surgery, either systemically or topically, to reduce excessive bleeding and transfusion requirements.

Other hemorrhagic conditions in which TXA has been shown effective are epistaxis, hemoptysis, endoscopic ear surgery, mastectomy, and hereditary hemorrhagic telangiectasia with bleeding.

For gastrointestinal bleeding, the effectiveness of TXA is controversial. Based on the most recent large randomized controlled trial, TXA is unlikely to confer additional benefit beyond the current standard of care in patients with severe upper or lower GI bleeding. However, this study had some limitations as most patients presented more than three hours after bleeding onset and a large portion were treated for presumed variceal bleeds.

According to some other studies, TXA use may be effective in reducing severe bleeding, blood transfusions, length of stay, and hospitalization costs, need for urgent endoscopy, the risk of re-bleeding, and the need for surgery. A recent meta-analysis revealed that TXA significantly reduced the rates of continued bleeding, urgent endoscopic intervention, and mortality compared to placebo.

Topical use of TXA may be more beneficial than systemic use as it may provide a higher drug concentration on the wound surface with negligible systemic concentrations. Most publications concerning topically administered TXA come from orthopedic literature where instilling TXA as a bolus into the joint reduces bleeding. Recently, a study revealed that intradermal injections of TXA in dermatological surgery reduces bleeding, especially in those on anticoagulant medications.

In gastroenterology practice, the topical use of TXA was investigated in one recent study which revealed that it conferred no additional benefit over standard care in patients with upper gastrointestinal hemorrhage.

In orthopedic patients, in addition to a reduction in bleeding, TXA was found to significantly improve postoperative pain.

While TXA is an inhibitor of fibrinolysis, and therefore might theoretically increase the risk of thrombotic vascular events, most studies show no increased risk of thromboembolism. This finding has been consistent with all routes of TXA administration including IV, topical/intra-articular, and other routes.

The investigators propose that the addition of TXA instead of adrenaline into the gel for injection during ER procedures may reduce intraprocedural and postprocedural bleeding, while also decreasing side effects of adrenaline injection including postprocedural pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for endoscopic resection of non-neoplastic and neoplastic lesions in the colon presenting to our tertiary academic center.
* Age > 18 years

Exclusion Criteria:

* patients with histories of allergic reactions to TXA
* history of seizures
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Postprocedural bleeding | Within 2 weeks of procedure
  Overt postprocedural bleeding, whether including a drop in hemoglobin or not

SECONDARY OUTCOMES:
Intraprocedural bleeding | During the procedure
  Bleeding during the procedure requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anton Bermont, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Technology Committee; Hwang JH, Konda V, Abu Dayyeh BK, Chauhan SS, Enestvedt BK, Fujii-Lau LL, Komanduri S, Maple JT, Murad FM, Pannala R, Thosani NC, Banerjee S. Endoscopic mucosal resection. Gastrointest Endosc. 2015 Aug;82(2):215-26. doi: 10.1016/j.gie.2015.05.001. Epub 2015 Jun 12. PMID 26077453
- [Background] Park CH, Lee SK. Preventing and controlling bleeding in gastric endoscopic submucosal dissection. Clin Endosc. 2013 Sep;46(5):456-62. doi: 10.5946/ce.2013.46.5.456. Epub 2013 Sep 30. PMID 24143302
- [Background] Fahrtash-Bahin F, Holt BA, Jayasekeran V, Williams SJ, Sonson R, Bourke MJ. Snare tip soft coagulation achieves effective and safe endoscopic hemostasis during wide-field endoscopic resection of large colonic lesions (with videos). Gastrointest Endosc. 2013 Jul;78(1):158-163.e1. doi: 10.1016/j.gie.2013.02.030. Epub 2013 Apr 6. PMID 23570622
- [Background] Lee HS, Jeon SW, Kwon YH, Nam SY, Shin S, Kim R, Ahn S. Prophylactic endoscopic coagulation to prevent delayed post-EMR bleeding in the colorectum: a prospective randomized controlled trial (with videos). Gastrointest Endosc. 2019 Nov;90(5):813-822. doi: 10.1016/j.gie.2019.05.039. Epub 2019 Jun 5. PMID 31175874
- [Background] Liaquat H, Rohn E, Rex DK. Prophylactic clip closure reduced the risk of delayed postpolypectomy hemorrhage: experience in 277 clipped large sessile or flat colorectal lesions and 247 control lesions. Gastrointest Endosc. 2013 Mar;77(3):401-7. doi: 10.1016/j.gie.2012.10.024. Epub 2013 Jan 11. PMID 23317580
- [Background] Castro R, Libanio D, Pita I, Dinis-Ribeiro M. Solutions for submucosal injection: What to choose and how to do it. World J Gastroenterol. 2019 Feb 21;25(7):777-788. doi: 10.3748/wjg.v25.i7.777. PMID 30809079
- [Background] Rex DK, Lahr RE, Peterson MM, Vemulapalli KC. Impact of including epinephrine in the submucosal injectate for colorectal EMR on postprocedural pain: a randomized controlled trial. Gastrointest Endosc. 2022 Mar;95(3):535-539.e1. doi: 10.1016/j.gie.2021.11.043. Epub 2021 Dec 9. PMID 34896443
- [Background] Cai J, Ribkoff J, Olson S, Raghunathan V, Al-Samkari H, DeLoughery TG, Shatzel JJ. The many roles of tranexamic acid: An overview of the clinical indications for TXA in medical and surgical patients. Eur J Haematol. 2020 Feb;104(2):79-87. doi: 10.1111/ejh.13348. Epub 2019 Dec 16. PMID 31729076
- [Background] Watts G. Utako Okamoto. Lancet. 2016 Jun 4;387(10035):2286. doi: 10.1016/s0140-6736(16)30697-3. No abstract available. PMID 27308678